CLINICAL TRIAL: NCT03576599
Title: Intravenous Bisphosphonate in Stress Fracture Treatment
Brief Title: Intravenous Bisphosphonate in Stress Fracture Treatment -A Randomised Controlled Double Blinded Multicenter Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficult to include patients
Sponsor: Oslo University Hospital (Other)
Collaborators: Betanien Hospital (Other); Sykehuset Ostfold (Other)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REK 2014/1986
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-07

CONDITIONS: Stress Fracture Foot; Stress Fracture Ankle
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoledronic Acid Injectable Product (Active Comparator): Patients randomized to treatment with Zoledronic Acid 5mg infusion, repeated after 3 months
  Interventions: Drug: Zoledronic Acid Injectable Product
- Placebo (Placebo Comparator): Patients randomized to Placebo infusion (saline), repeated after 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid Injectable Product — One Group are randomiced to Zoledronic Acid Injectable Product and one Group to Placebo
  Other Names: Aclasta
  Arms: Zoledronic Acid Injectable Product
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The effect of an intravenous bisphosphonate (zoledronic acid) on healing and symptoms of stress fractures that do not respond to conservative/conventional treatment within 6 months, will be investigated.

DETAILED DESCRIPTION:
Randomised controlled multicenter trial. Prospective study. The trial will be performed in accordance with the CONSORT-statement. The inclusion period will be two years. The patients will be randomised to standard treatment (casting, partial weight-bearing, orthotic insoles) in addition to either zoledronic acid or placebo (saline) infusions. The randomization process will be carried out through a web based randomization service (Norwegian University of Science and Technology, Unit for applied clinical research). Patient data will be kept and organized by a study coordinator (nurse) and will not be revealed for the clincal investigators, except in medical emergency situations. In such cases, the patient will be excluded from the study. A number of bottles containing zoledronic acid or placebo will be available in each of the participating hospitals. The bottles containing zoledronic acid and placebo are visually identical, numbered from 1 through 80 (two bottles with similar number, the second bottle will be kept for the second infusion). The patients will be randomised in blocks, creating evenly sized groups given zoledronic acid or placebo. When a patient is included and thereafter randomised, the study coordinator decides which bottle number to be given and provides this information to the physician. The study coordinator is the only person in the study group which is not blinded.

On the first visit, the included patients will undergo clinical examination and baseline parameters will be registered. If MRI is not previously obtained, this will be performed as quickly as possible. The clinical controls will be scheduled 4 and 12 and 26 weeks thereafter, the latter including MRI. If healing has still not occured, the patients will be given the second infusion and meet for clinical examination every 4 weeks until healing. Clinical healing is defined as painless or near painless (VAS pain 0-2) weight bearing. If healing has not occured 12 months after inclusion, surgery will be considered.

MRI will be obtained at (or before) baseline, 6 months and one year. MRIs will be examined by a blinded radiologist. Bone marrow lesions (BMLs) will be measured (area and volume) and fracture lines registered.

All patients (both groups) will be prescribed calcium and vitamin D (Calcigran Forte 500mg/400IE) taken orally once daily in the whole study period. This is recommended as an adjunct to bisphosphonate treatment on a general basis/standard treatment and is not to be investigated separately.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Stress fractures in the foot. A stress fracture is defined as a fracture occured after repetitive trauma, with characteristic MRI findings (ref) and distinctive pain over the fracture site at weight bearing.
* at least 6 months of pain history
* compliant patient
* non-aided ambulatory patient prior to the injury

Exclusion Criteria:

* Ongoing use of bisphosphonates, PTH/PTH-analogues or use within 12 months prior to the injury
* Use of bisphophonates for more than 6 months within the last 5 years
* Intolerance to zoledronic acid
* Renal failure (GFR<30)
* S-25(OH)vitD > 25
* pregnancy
* breast feeding
* hypocalcemia
* MRI contraindications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
The American Orthopedic Foot and Ankle Score (AOFAS) mid foot scale | 1 year
  a scale evaluating pain, function and alignment of the foot. 0-100, With 100 as maximum score

SECONDARY OUTCOMES:
Visual analoge scale (VAS) for pain | 3, 6, 8, 10 and 12 months
  Patient Reported Outcome Measure (PROM) for evaluating local pain
Change in bone marrow lesions evaluated by magnetic resonance imaging (MRI) | 1 year
  the intensity and the amount of bone marrow oedema is evaluated
The American Orthopedic Foot and Ankle Score (AOFAS) mid foot scale | 3, 6, 8, 10, 12 months
  a scale evaluating pain, function and alignment of the foot

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth E Husebye, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway